CLINICAL TRIAL: NCT06127862
Title: The Effect of Environmental Health Education on Microplastica Pollution Awareness
Brief Title: Microplastica Pollution Awareness Level of Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, FATOŞ UNCU, ASSISTANT PROFESSOR, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FU-PHN-FU-01
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Environmental-Pollution-Related Condition
Keywords: Enviromental health; Microplastics; Student

STUDY DESIGN:
Intervention Model Description: This research is a randomised control study with pretest-posttest design.
Who Masked: Participant
Masking Description: Participants were assigned to the groups by a single-blind design. For allocation, intervention and control groups were coded as "A" and "B". Which letter would be the intervention or control group was determined by the coin toss method before the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Other): The forms used in the study were collected by the researcher through face-to-face interviews in seminar halls in schools. First of all, students in the experimental group were educated about environmental health and microplastica, and nursing interventions were made. The training was organized for twenty minutes in each session, with a total of four sessions at two-week intervals. Personal Information Form and Microplastica Pollution Awareness Scale (MPAS) were filled out as a pre-test in the seminar halls of the schools under the supervision of the researcher.
  Interventions: Other: Education group
- Control group (Other): Personal information form and Microplastica Pollution Awareness Scale (MPAS)" were applied to the students in the control group as a pre-test. No training was given to the control group. Fifteen days after the end of the fourth training of the intervention group, the MPAS was applied to the control group as a post-test, and data collection was terminated. After the post-test was administered to the groups, training materials were also given to individuals from the control group who requested them.
  Interventions: Other: No training was given

INTERVENTIONS:
Other: Education group — Students in the experimental group were educated about environmental health and microplastica, and nursing interventions were made. The training was organized for twenty minutes in each session, with a total of four sessions at two-week intervals.
  Arms: Education group
Other: No training was given — No training was given
  Arms: Control group

SUMMARY:
This study aims to raise awareness among individuals about plastic and microplastica pollution, reduce plastic consumption, reduce the amount of plastic waste that grows cumulatively every year, and contribute to the development of a livable environment.

DETAILED DESCRIPTION:
The aim of this research is to investigate the effect of environmental health education given at the 9th-grade level on the microplastica pollution awareness level of students.

This pretest-posttest experimental study with a randomized control group was conducted between 2022 and 2023 in three high schools in a province in eastern Turkey. The sample of the study consisted of 90 ninth-grade students (experimental group: 45, control group: 45), and the sample magnitude was determined by power analysis. Tools such as the "Personal Information Form" and "Microplastica Pollution Awareness Scale (MPAS)" were used to collect data. Training was given to the experimental group as a nursing intervention in a total of 4 sessions at 15-day intervals. No intervention was applied to the individuals in the control group. In the data evaluation process, percentage distribution, arithmetic mean, standard deviation, chi-square test, correlation and regression analyses were used.

While no significant difference was observed in the MPAS total score in the control group according to the pre-test and post-test mean scores, a significant difference was observed in the MPAS total score in the experimental group (p≤0.05). When the posttest mean scores of the experimental and control groups were examined, it was observed that the posttest mean scores of the experimental group were higher than the posttest mean scores of the control group and there was a statistically significant difference (p≤0.05).

It was observed that the microplastica pollution awareness level of the experimental group students who received environmental health training increased significantly.

ELIGIBILITY:
Inclusion Criteria:

* age group of 13-15 years,
* 9th-grade students,
* without any intellectual disability,
* with parental consent.

Exclusion Criteria:

* Previous or current participation in an MPAS training,
* Inability to obtain parental consent.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Microplastica Pollution Awareness Scale | 3 MONTHS
  MPAS has a 3-factor structure. It consists of 5 negative and 9 positive items. The questions were prepared to measure the level of awareness of microplastica pollution. The Likert scale consists of 1 point= "no", 2 points= "not sure" and 3 points= "yes" options. The highest score that can be obtained from the scale is 42 points. The increase in the score obtained from the scale is consistent with the participant's awareness of microplastica pollution

CONTACTS AND LOCATIONS:
Overall Officials: FATOŞ UNCU, PhD, Principal Investigator — Firat University
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No